CLINICAL TRIAL: NCT04361201
Title: Analysis of the Ligamentization Process in the Anatomical Ligamentoplasty of the Lateral Ankle Plane to the Hamstrings
Acronym: LIGANALYS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200788; 2020-A01317-32 (Registry Identifier: IDRCB)
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2022-04

CONDITIONS: Ligament Plastic Surgery
Keywords: ligament injury; ligamentization
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ligament plastic surgery ankle: Patient treated priorly by ligament plastic surgery of lateral ankle plane under arthroscopy
  Interventions: Procedure: Ligament plastic surgery; Diagnostic Test: RMI and ultrasound
- Control group: Controlateral ankle
  Interventions: Procedure: Ligament plastic surgery; Diagnostic Test: RMI and ultrasound

INTERVENTIONS:
Procedure: Ligament plastic surgery — Ligament plastic surgery of ankle under arthroscopy for recurrent instable ankle reason and failure of medical treatment.
Diagnostic Test: RMI and ultrasound — RMI examination at 3 months on operated ankle, and 3 CT scan examinations with elastography module will be performed at planned timeframes.

SUMMARY:
This is a prospective bi-centric study, which evaluate the evolution of RMI signal of transplant till 12 months after ligament plasty surgery.

As the primary objective, the study aims to define the post-operative timeframe needed to obtain an optimal quality of repair, especially in their restarting of sportive activities, by analysis of RMI signal and biomechanic features modifications.

As secondary objectives, the study aims to:

* study the correlation between the RMI signal of plasty and the Young's modulus;
* study the evolution of RMI of plasty at M3, M6 and M12;
* study the evolution of Young's modulus at M3, M6 and M12;
* evaluate the reproductibility between 2 lector of RMI measurements;
* evaluate the reproductibility between 2 lector of elastography measurements of LTFA;
* evaluate the optimal delay of return to sport after ligament plasty surgery of ankle;
* develope a score of type SNQ for ankle ligament plasty surgery;
* evolution of AOFAS and EVA scores.

DETAILED DESCRIPTION:
The eligible patients will be enrolled in the department of orthopaedic surgery of Ambroise Paré hospital, each patient will undergo a 12-months follow-up in the department of orthopaedic surgery in Armand Trousseau hospital for the elastography evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated priorly by ligament plastic surgery of lateral ankle plane under arthroscopy;
* Affiliated to or covered by the French social security - welfare system in France;
* Have provided written informed consent for the study;
* Be >/= 18 years of age on day of signing informed consent.

Exclusion Criteria:

* Patients who undergo iterative surgery or have history of contralateral surgery;
* Patient under guardianship or curatorship;
* Unable to understand the proposed study or provide written informed consent for the study;
* Foreign patients under AME schema, a medical help from the state in France;
* Pregnant or breastfeeding woman;
* Patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent a ligament plastic surgery of lateral ankle plane under arthroscopy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Classification of RMI signal | At 3 months
  The classification of RMI signal will be defined as:
  * frank hyposignal: stage 1;
  * intermediary signal (close to muscles of T2): stage 2;
  * moderate hypersignal (close to cartilage of T2): stage 3;
  * intensive hypersignal (close tointra-articular liquid of T2): stage 4.
Classification of RMI signal | At 6 months
  The classification of RMI signal will be defined as:
  * frank hyposignal: stage 1;
  * intermediary signal (close to muscles of T2): stage 2;
  * moderate hypersignal (close to cartilage of T2): stage 3;
  * intensive hypersignal (close tointra-articular liquid of T2): stage 4.
Classification of RMI signal | At 12 months
  The classification of RMI signal will be defined as:
  * frank hyposignal: stage 1;
  * intermediary signal (close to muscles of T2): stage 2;
  * moderate hypersignal (close to cartilage of T2): stage 3;
  * intensive hypersignal (close tointra-articular liquid of T2): stage 4.

SECONDARY OUTCOMES:
Anterior talofibular ligament measurement | At 3, 6 and 12 months
  anterior talofibular ligament measurement will be performed by RMI
Calcaneofibular ligament measurement | At 3, 6 and 12 months
  calcaneofibular ligament measurement will be performed by RMI
Elastography | At 3, 6 and 12 months
  Elastography measurements: Young's Modulu
Pain evaluation | At baseline and 3, 6 and 12 months
  By the American Orthopedic Foot and Ankle Score (AOFAS) to evaluate the pain.
Pain evaluation | At baseline and 3, 6 and 12 months
  By the visual analog scale (VAS) to evaluate the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre HARDY, MD, Principal Investigator — Orthopaedic Surgery Department, Ambroise Paré hospital, APHP; Thomas BAUER, MD, Study Director — Orthopaedic Surgery Department, Ambroise Paré hospital, APHP
Locations (1):
- Orthopaedic Surgery Department, Ambroise Paré hospital, APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No